CLINICAL TRIAL: NCT06655883
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Suvorexant for the Treatment of Insomnia in Participants With Opioid Use Disorder
Brief Title: A Study of Suvorexant (MK-4305) for the Treatment of Insomnia Disorder in Participants With Opioid Use Disorder (MK-4305-098)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4305-098; MK-4305-098 (Other: MSD)
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Suvorexant (Experimental): Participants receive 10 mg of suvorexant for the first three nights, increased to 20 mg of suvorexant nightly thereafter at the investigator's discretion, for up to approximately 8 weeks.
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Participants receive suvorexant-matching placebo for up to approximately 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Oral Tablet
  Other Names: MK-4305
  Arms: Suvorexant
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
People with opioid use disorder (OUD) can have trouble falling or staying asleep. Researchers want to know if suvorexant will help people with OUD fall asleep and stay asleep. The goal of this study is to learn about the safety of suvorexant and how well people tolerate it. Researchers also want to learn if suvorexant helps people sleep longer compared to people who take placebo. A placebo looks like the study medicine but has no actual study medicine in it.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a primary diagnosis of OUD according to Diagnostic and Statistical Manual of Mental Disorder, 5th Edition (DSM-5), and confirmed through the Mini International Neuropsychiatric Interview (MINI).
* Is on a verified, stable dose of medications for opioid use disorder (MOUD) treatment.
* Meets DSM-5 criteria for the diagnosis of Insomnia Disorder
* Has a regular bedtime between 8 PM (20:00) and 1 AM (01:00) and is willing to maintain it for the duration of the study.
* Has not used opioids for a period of at least 4 weeks before entering the study.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has current uncontrolled major co-morbid psychiatric illness including major depressive disorder, bipolar disorder, schizophrenia, or any psychiatric condition with psychotic features.
* Has current diagnosis or history within 5 years of any of the following: narcolepsy, sleep paralysis, severe periodic limb movement disorder, restless leg syndrome, cataplexy, circadian rhythm sleep disorder, parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, rapid eye movement (REM) behavior disorder, significant degree of sleep-related breathing disorder, excessive daytime sleepiness (EDS), or primary hypersomnia.
* Is at imminent risk of self-harm.
* Has a known history of stroke that may confound the diagnosis of insomnia.
* Has a clinically significant movement disorder such as akinesia.
* Has a history of hepatitis or live disease.
* Has habitual use of central nervous system (CNS)-depressants or stimulants that may be responsible for the participant's disturbed sleep.
* Has a history of malignancy, ≤3 years prior to start of study, with the exception of nonmelanoma skin cancer, prostate cancer or localized carcinoma in situ of the cervix.
* Has a history of hypersensitivity to more than 3 chemical classes of drugs, including prescription and over-the-counter medications.
* Has donated blood products or had phlebotomy within 8 weeks prior to start of study.
* Has a history of transmeridian travel within 2 weeks prior to start of study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-06-24 (Estimated); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Sleep Time at Week 8 | Baseline and Week 8
  Total sleep time will be measured in a sleep laboratory by polysomnography at the participant's habitual bedtime. Change from baseline in total sleep time at Week 8 will be reported.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 10 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Experience One or More Serious Adverse Events (SAEs) | Up to approximately 10 weeks
  An SAE is any untoward medical occurrence that at any dose results in death, is life threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect or is another important medical event deemed such by medical or scientific judgement.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Change from Baseline in Wakefulness after Persistent Sleep Onset at Week 8 | Baseline and Week 8
  Wakefulness after persistent sleep onset will be measured in a sleep laboratory by polysomnography at the participant's habitual bedtime. Change from baseline in wakefulness after persistent sleep onset at Week 8 will be reported.
Number of Participants Who are Positive for Substance Abuse at Day 1 | Day 1
  A positive assessment for substance abuse at Day 1 is defined as either a positive urine drug test for opioids and other nonmedical substances including fentanyl, cocaine, amphetamines, benzodiazepines, and cannabis OR a positive response on the Substance Use History (SUH) Since Last Assessment questionnaire. The Substance Use History Questionnaire (SUH) has been developed specifically for this study. This is a self-reported questionnaire used to obtain a variety of quantitative estimates of cannabis, alcohol, and other nonmedical substance use. The SUH Since Last Assessment Questionnaire will be used to assess nonmedical substance and alcohol use since the previous study visit.
Number of Participants Who are Positive for Substance Abuse at Day 4 | Day 4
  A positive assessment for substance abuse at Day 4 is defined as either a positive urine drug test for opioids and other nonmedical substances including fentanyl, cocaine, amphetamines, benzodiazepines, and cannabis OR a positive response on the Substance Use History (SUH) Since Last Assessment questionnaire. The Substance Use History Questionnaire (SUH) has been developed specifically for this study. This is a self-reported questionnaire used to obtain a variety of quantitative estimates of cannabis, alcohol, and other nonmedical substance use. The SUH Since Last Assessment Questionnaire will be used to assess nonmedical substance and alcohol use since the previous study visit.
Number of Participants Who are Positive for Substance Abuse at Week 2 | Week 2
  A positive assessment for substance abuse at Week 2 is defined as either a positive urine drug test for opioids and other nonmedical substances including fentanyl, cocaine, amphetamines, benzodiazepines, and cannabis OR a positive response on the Substance Use History (SUH) Since Last Assessment questionnaire. The Substance Use History Questionnaire (SUH) has been developed specifically for this study. This is a self-reported questionnaire used to obtain a variety of quantitative estimates of cannabis, alcohol, and other nonmedical substance use. The SUH Since Last Assessment Questionnaire will be used to assess nonmedical substance and alcohol use since the previous study visit.
Number of Participants Who are Positive for Substance Abuse at Week 4 | Week 4
  A positive assessment for substance abuse at Week 4 is defined as either a positive urine drug test for opioids and other nonmedical substances including fentanyl, cocaine, amphetamines, benzodiazepines, and cannabis OR a positive response on the Substance Use History (SUH) Since Last Assessment questionnaire. The Substance Use History Questionnaire (SUH) has been developed specifically for this study. This is a self-reported questionnaire used to obtain a variety of quantitative estimates of cannabis, alcohol, and other nonmedical substance use. The SUH Since Last Assessment Questionnaire will be used to assess nonmedical substance and alcohol use since the previous study visit.
Number of Participants Who are Positive for Substance Abuse at Week 8 | Week 8
  A positive assessment for substance abuse at Week 8 is defined as either a positive urine drug test for opioids and other nonmedical substances including fentanyl, cocaine, amphetamines, benzodiazepines, and cannabis OR a positive response on the Substance Use History (SUH) Since Last Assessment questionnaire. The Substance Use History Questionnaire (SUH) has been developed specifically for this study. This is a self-reported questionnaire used to obtain a variety of quantitative estimates of cannabis, alcohol, and other nonmedical substance use. The SUH Since Last Assessment Questionnaire will be used to assess nonmedical substance and alcohol use since the previous study visit.
Number of Participants with Positive Urine Drug Screen | Day 1, Day 4, Week 2, Week 4, Week 8
  A positive urine drug screen is defined as urine drug test positive for opioids and other nonmedical substances including fentanyl, cocaine, amphetamines, benzodiazepines, and cannabis

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Johns Hopkins University ( Site 1001), Baltimore, Maryland
  - Medical University of South Carolina ( Site 1005), Charleston, South Carolina
  - Adams Clinical Dallas ( Site 2007), DeSoto, Texas
  - Memorial Hermann Village ( Site 2001), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com